CLINICAL TRIAL: NCT05706194
Title: Early Neurological Prognostication of Outcome After Out-of-hospital Cardiac arrest-a STEPCARE Prospective Substudy
Brief Title: Early Neuroprognostication After OHCA
Status: Recruiting | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Helsingborgs Hospital (Other); University of Helsinki (Other); Skane University Hospital (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: STEPCARE EARLY-NEURO
Record Dates: First submitted 2023-01-09; First posted 2023-01-31 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Arrest; Neurological Outcome; EEG; CT; Brain Injuries; Biomarkers
MeSH Terms: conditions — Heart Arrest; Brain Injuries | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Early neurological prognostication with biomarkers, EEG and CT — Biomarker samples collected at 12, 24, 48 and 72 h after randomisation, CT and EEG performed as early as possible after 24 h post randomisation in patients still unconscious (defined as not awake and able to follow verbal commands)

SUMMARY:
This is a prospective observational substudy of the STEPCARE trial ClinicalTrials.gov Identifier: NCT05564754) with the aim to examine whether prognostication of neurological outcome after cardiac arrest can be performed earlier than the 72 h time-point recommended by guidelines today.

DETAILED DESCRIPTION:
Hypotheses

1. The combination of clinical examination, the brain injury marker neurofilament light (NFL), electroencephalography (EEG), and head computed tomography (CT) predicts poor functional outcome already at 24 h post-arrest without false positive predictions.
2. Any guideline recommended method (EEG/CT/SSEP/clinical examination) fulfilling criteria for a poor outcome will have highly elevated blood levels of NFL, indicating the presence of severe brain injury.
3. Extensive sedation will not affect the prognostic accuracy of our prognostic methods EEG, NFL and CT.

Material and methods

The STEPCARE trial The patient population is adult patients with an out-of-hospital cardiac arrest with a presumed cardiac or unknown cause of arrest randomised in the STEPCARE trial (Sedation, TEmperature and Pressure after out-of-hospital Cardiac Arrest and REsuscitation, ClinicalTrials.gov Identifier: NCT05564754). The STEPCARE trial is an investigator initiated 2x2x2 international multicentre trial which will randomise patients to three intensive care interventions: minimal or higher levels of sedation, fever treatment versus no fever treatment and two different blood pressure targets. The aim of STEPCARE is to examine whether the interventions improves survival or functional outcome after CA. The statistical calculations indicate that 3500 patients are required to obtain sufficient power for our research questions. Patients will be recruited from more than 80 hospitals who have participated in the previous cardiac arrest trials initiated by the Lund University Center for Cardiac Arrest namely the TTM- and TTM2-trials (the to date largest published cardiac arrest trials).

The STEPCARE EARLY-NEURO substudy We will prospectively recruit participating sites who commit to follow the study protocol for participation in the biobank, and routinely examine patients' unconscious at 24 hours with EEG and CT as early as possible after 24 h. Serum and plasma blood samples will be collected prospectively at 12 h, 24 h, 48 h and 72 h post-randomisation, processed on site and transported to the Integrated Biobank in Luxembourg for storage. Biochemical analyses of NFL will be performed in batch after trial completion. The original EEG recordings, SSEP and neuroimaging (CT and MRI) will be collected for central blinded evaluation by study investigators. All patient data will be stored using patients study ID as identification. All patients will be treated according to the STEPCARE trial protocol according to randomisation, treatment, and follow-up. Prediction of neurological outcome performed according to the ERC/ESICM guidelines ≥72 hours post-arrest. Decisions on withdrawal of life-sustaining therapy will not be based on the early examinations alone, but must follow ERC/ESICM recommendations. Functional outcome will be assessed at a face-to-face follow up after six months and classified according to the modified Rankin Scale (mRS). Poor functional outcome will be defined as mRS 4-6 (moderately severe disability, severe disability, or death).

ELIGIBILITY:
Inclusion Criteria:

Adult cardiac arrest patients with an out-of-hospital cardiac arrest of non-traumatic cause treated at hospitals recruiting patients to the STEPCARE neuroprognostication substudy. Other inclusion criteria include:

* a minimum of 20 minutes without chest compressions
* Unconsciousness defined as not being able to obey verbal commands (FOUR-score motor response of <4) or being intubated and sedated because of agitation after sustained ROSC
* Eligible for intensive care without restrictions or limitations
* Inclusion within 4 hours of ROSC

Exclusion Criteria:

* On ECMO prior to randomisation
* Pregnancy
* Suspected or confirmed intracranial hemorrhage
* Previously randomised in the STEPCARE trial
* Patients with limitations in level-of-care due to for example generalized malignancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac arrest patients with an out-of-hospital cardiac arrest of any non-traumatic cause treated at hospitals recruiting patients to the STEPCARE neuroprognostication substudy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | Six months post-randomisation
  Poor outcome defined as modified Rankin Scale 4-6

SECONDARY OUTCOMES:
Blood levels of brain injury markers | Samples collected at 12-72 hours post-randomisation
  Neurofilament light

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Nielsen, MD, PhD, Study Chair — Lund University
Locations (4):
- Helsinki Hospital, Helsinki, Finland
- Charité University Hospital, Berlin, Germany
- Sweden (2):
  - Helsingborgs Hospital, Helsingborg
  - Skane University Hospital, Lund

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request following publication

DOCUMENTS (1):
  • Study Protocol (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT05706194/Prot_000.pdf